CLINICAL TRIAL: NCT01162980
Title: The ACEi SwitchBack Study
Brief Title: The Angiotensin Converting Enzyme (ACE) Inhibitor SwitchBack Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Servier (Industry)
Responsible Party: Dr Nadia Giannetti, McGill University Health Centre
Other Study IDs: 09-150-BMB (SWITCHBACK)
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-07

CONDITIONS: Heart Failure
Keywords: ACE inhibitors; ARBs
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
ACE inhibitors have been studied extensively in the treatment of heart failure and have been shown to be beneficial in all its stages. Studies with the use of angiotensin receptor blockers (ARBs) in chronic heart failure have not shown equivalent results. Many patients are on an ARB for a variety of reasons. Some of these may have had cough as a symptom of heart failure and not due to medication side effect. According to guidelines, angiotensin converting enzyme inhibitors (ACEi) are still first-line therapy in the treatment of heart failure. As ACEi have been extensively studied showing improvement in morbidity and mortality all patients should be on this treatment unless absolutely contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* heart failure patients who have indications for ACEi but are currently on ARBs with no absolute contraindications to ACEi
* patients with an ejection fraction of < or = 35% verified in the last 12 months by echo, angio, or nuc med who are NYHA class I to IV and followed in a heart failure clinic for three months
* on beta-blockers, unless contra-indicated
* stable on current meds for 3 months (except dose of diuretics)
* able to give informed consent

Exclusion Criteria:

* documented angioedema/anaphylaxis with prior ACEi use
* documented worsening renal failure, hyperkalemia, cough and gastrointestinal symptoms that are definitely believed to be due to ACEi
* potassium >5.0 mmol/L

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: heart failure patients followed in heart failure clinics in Canada
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-01 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
proportion of patients on ARB who are switched back to ACEi and\ who tolerate ACEi | 6 months
  Patients with heart failure who are on ARB who do not clear contra-indication to ACEi will be switched to an ACei. their tolrance to this will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Giannetti, MD, Principal Investigator — Royal Victoria Hospital, McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada